CLINICAL TRIAL: NCT06733558
Title: Long-term Potentiation Disruption Underlying Cognitive Impairment in ECT
Acronym: LTP-DUCIECT
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: NIGMS, the funding agency, does not consider this study a clinical trial and they asked to remove from the system.
Sponsor: University of New Mexico (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-286; 5P20GM109089-10 (NIH)
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder; Bipolar Disorder II
Keywords: electroconvulsive therapy; brain recovery; major depressive disorder; long-term potentiation; cognitive impairment; bipolar disorder, type II
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Cognitive Dysfunction | interventions — Electroconvulsive Therapy

STUDY DESIGN:
Intervention Model Description: There will be only one group that will be studied, those undergoing ECT.
Masking Description: Masking will not be necessary, as there is only one group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants undergoing ECT (Experimental): Participants undergoing ECT for depressive episode
  Interventions: Procedure: Electroconvulsive Therapy

INTERVENTIONS:
Procedure: Electroconvulsive Therapy — Electroconvulsive therapy (ECT) is a medical treatment that uses controlled electrical stimulation to induce a brief, generalized seizure in the brain. This intervention is performed under general anesthesia with muscle relaxants to ensure patient comfort and safety. ECT is typically used to treat severe depression, bipolar disorder, and other mental health conditions when other treatments, such as medication and psychotherapy, have not been effective.

SUMMARY:
Cognitive problems, like memory loss, are common after brain injuries like trauma or stroke. These problems make daily life harder, and the investigators don't yet know the best ways to help the brain recover. Scientists think that a process in the brain called long-term potentiation (LTP) is important for memory and learning. When LTP isn't working properly, it may cause problems with thinking and memory. But studying LTP in people is hard because it happens deep inside the brain.

Our research uses a treatment called electroconvulsive therapy (ECT) to better understand LTP. ECT is a treatment for severe depression that works by causing a controlled seizure in the brain. While ECT often helps depression, it can temporarily cause memory and thinking problems, which usually improve over time. This makes ECT a good way to study how thinking and memory recover.

The investigators will use a tool called electroencephalography (EEG) to measure brain activity during different stages of ECT treatment. EEG is a safe and non-invasive way to track changes in LTP. Specifically, the investigators will measure how the brain responds to visual signals using something called visual evoked potentials (VEPs). These signals can show how LTP is affected by ECT.

The study's main goal is to track changes in LTP using VEPs during and after ECT. By studying these changes, the investigators hope to learn how ECT affects the brain and how it recovers. This could help improve treatments for brain injuries and other conditions that cause memory and thinking problems.

DETAILED DESCRIPTION:
This study aims to investigate changes in long-term potentiation (LTP)-like phenomena using visual evoked potentials (VEPs) in patients undergoing electroconvulsive therapy (ECT) for treatment-resistant depression. LTP is a fundamental neurophysiological process involved in synaptic plasticity and memory formation, and its disruption has been proposed as a potential mechanism underlying the cognitive side effects of ECT.

Study Design:

The study employs a paired pre- and post-intervention design. VEPs will be recorded using electroencephalography (EEG) at two time points:

Pre-ECT: Prior to the initiation of the ECT treatment series. Post-ECT: Immediately following the completion of the ECT series. The VEP paradigm consists of repetitive visual stimulation presented on a computer monitor. The primary outcome is the amplitude of the N1 component of the VEP, a negative deflection occurring approximately 100 milliseconds after stimulus onset, which is sensitive to changes in LTP-like synaptic plasticity.

Methodology:

Participants will undergo EEG sessions using a high-density EEG system with either a 64-lead cap. Visual stimuli will be presented in a controlled environment to elicit VEPs, and the data will be analyzed to assess changes in the N1 component amplitude between the pre- and post-ECT recordings.

Analysis:

A paired t-test will be used to compare N1 amplitudes before and after the ECT series to evaluate the hypothesis that ECT disrupts LTP-like phenomena, as reflected by changes in VEPs.

This study provides a novel application of VEPs to investigate the neurophysiological effects of ECT and aims to enhance our understanding of synaptic plasticity in the context of therapeutic brain stimulation. Findings from this research could inform future strategies to mitigate the side effects of ECT while preserving its clinical efficacy.

ELIGIBILITY:
Inclusion criteria:

* diagnosis of major depressive disorder (MDD; with or without psychotic features) or bipolar 2 most recent episode depressed;
* clinical indications for ECT with right unilateral electrode placement including treatment resistance or a need for a rapid and definitive response,
* age range adults 18-85 years, and
* English-speaking (many of the neuropsychological tests are only available in English). Antidepressant medications will be continued as clinically indicated. To maintain feasibility and retention, as needed medications will be permitted for anxiety and insomnia.

Exclusion criteria:

* Defined neurological or neurodegenerative disorder (e.g., traumatic brain injury, epilepsy, Alzheimer's disease);
* other psychiatric conditions (e.g., schizophrenia, bipolar I disorder);
* current drug or alcohol use disorder (except for nicotine);
* prisoners; and
* pregnancy (pre- menopausal participants will receive pregnancy test, which is clinically indicated for ECT and not part of study protocol).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-21 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Visual Evoked Potential | From enrollment to eight weeks after enrollment
  The primary outcome of this study is to measure changes in long-term potentiation (LTP)-like phenomena using visual evoked potentials (VEPs), a non-invasive marker of brain activity recorded through electroencephalography (EEG). VEPs are brain responses to visual stimuli, and the N1 component, a negative peak occurring approximately 100 milliseconds after the stimulus, serves as a reliable index of LTP-like phenomena in humans.
  In this study, participants will undergo a visual stimulation paradigm designed to elicit and measure changes in the amplitude of the N1 component. This approach allows us to assess changes in synaptic plasticity (a key feature of LTP) before, during, and after a series of electroconvulsive therapy (ECT) treatments. These measurements will be correlated with cognitive performance and memory changes to explore the relationship between ECT-induced cognitive effects and LTP disruption.

CONTACTS AND LOCATIONS:
Locations (1):
- Domenici Hall, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share individual participant data (IPD) is currently undecided. While the study aims to contribute to scientific knowledge and improve understanding of electroconvulsive therapy (ECT)-associated cognitive impairment, logistical and regulatory considerations regarding data de-identification, storage, and sharing policies are still under review. The research team is evaluating whether sharing IPD, such as de-identified EEG data and cognitive performance results, would align with institutional guidelines and participant consent. Updates on the IPD sharing decision will be provided upon final determination.